CLINICAL TRIAL: NCT07266506
Title: Development of an Eating Behavior Risk Score
Acronym: PACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Professor, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00023903
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Childhood
Keywords: Obesity; Eating Behaviors; Appetite Regulation; Functional magnetic resonance imaging; Food-cue reactivity
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children in PACE Phenotype Study (Experimental): A total of 210 child-parent dyads (420 participants total) will be followed for 12 months to investigate the neurobiological and behavioral aspects of the PACE eating phenotype and its relationship to adiposity in children. Children will be 7 to 9 years old, with a body mass index (BMI)-for-age percentile either below the 85th or at or above the 95th percentile. The biological mother will have a BMI categorized as either normal weight (18.5-25.0 kg/m²) or obese (≥30.0 kg/m²). The study will assess brain responses to food cues, eating behaviors, and body fat using DXA scans, along with family socioeconomic and feeding factors that may influence weight gain trajectories.
  Interventions: Behavioral: Assessment of PACE Eating Phenotype and Related Behavioral and Neurobiological Measures

INTERVENTIONS:
Behavioral: Assessment of PACE Eating Phenotype and Related Behavioral and Neurobiological Measures — This study does not involve an active intervention. The exposures of interest include the children's eating behaviors as measured by the PACE phenotype score, which encompasses portion size responsiveness, appetite traits, loss of control eating, and eating rate. Brain responses to food cues assessed by fMRI, body composition measured by DXA, and family socioeconomic status will also be evaluated as key exposures. These measures will be collected at baseline and at 12-month follow-up to examine associations with adiposity and behavioral outcomes.

SUMMARY:
This study will explore how children's eating behaviors are connected to brain activity and body fat levels. Researchers are especially interested in a behavior pattern called the PACE phenotype, which includes how much children eat when offered large portions, how quickly they eat, their appetite traits, and their ability to control eating. The goal is to better understand why some children are more likely to gain weight than others.

The study will include children between the ages of 7 and 9 and will follow them for one year. Researchers will use brain scans, lab-based meal observations, and questionnaires to study how children respond to food and how their eating patterns relate to body fat at the start of the study and one year later. The study will also look at how family background, parenting, and other factors might protect some children from gaining excess weight even if they show risky eating behaviors. Results may help identify which children are most at risk for obesity and guide future strategies for prevention.

DETAILED DESCRIPTION:
This is a one-year observational study designed to better understand how certain eating behaviors in children relate to brain function and weight gain over time. These behaviors will be assessed using a combination of laboratory meal tasks, caregiver questionnaires, and behavioral coding. Children will be invited to six research visits-four at the beginning of the study and two 12 months later-during which they will participate in structured meals where portion sizes are adjusted, complete computer-based and paper assessments, and undergo brain imaging while viewing pictures of food. Body composition will be measured at both timepoints using a DXA scan. In addition, researchers will collect information on children's sleep, physical activity, executive function, dietary intake, and interoceptive awareness. Parents will be asked to complete surveys about their family's socioeconomic background, food security, feeding practices, and their child's behavior, temperament, and development. One of the study's goals is to examine how brain regions involved in appetite regulation and self-control respond to food cues in children with different PACE scores. Another goal is to determine whether children with higher PACE scores tend to have more body fat and whether those scores predict changes in body fat over one year. The study will also explore whether children from families with higher or lower socioeconomic status show different patterns of risk. Finally, researchers will use a machine learning approach to identify children who seem resilient to weight gain, despite having high-risk eating patterns, and to better understand what family or individual characteristics might explain that resilience.

ELIGIBILITY:
Inclusion Criteria:

Children :

* Children must be of good health (with the exception of obesity being allowed) based on parental self-report.
* Children should have no learning disabilities or developmental delays (e.g., ADHD, Autism, dyslexia)
* Children should speak English fluently.
* Children should not be on any medications known to influence body weight, taste, food intake, behavior, or blood flow, not be claustrophobic.
* Children should between the ages of 7-9 years-old at enrollment.
* Children must have a BMI-for-age % < 85 or ≥ 95 to be enrolled.
* The biological mother must have a BMI between 18.5 - 25.0 kg/m2 or a BMI ≥ 30.0 kg/m2. The parent primarily in charge of feeding must be able to accompany children to the visits.

Parents :

* The biological mother must have a BMI between 18.5 - 25.0 kg/m2 or a BMI ≥ 30.0 kg/m2. The parent primarily in charge of feeding must be able to accompany children to the visits.
* The parent who has the most knowledge of the child's eating behavior, media access, sleep and behavior must be available to attend the visits with their child. This would be decided among the parents.

Exclusion Criteria:

Children :

* They are not within the age requirements (< 7 years-old or > 9 years-old) at baseline.
* They are taking cold or allergy medication, or other medications known to influence cognitive function, taste, appetite, or blood flow.
* They are red/green colorblind.
* They do not speak English fluently.
* They report being claustrophobic, or if they have any of the following: a learning disability, ADD/ADHD, language delays, autism, dyslexia, a pre-existing medical condition such as type I or type II diabetes, rheumatoid arthritis, Cushing's syndrome, Down's syndrome, food allergies, severe lactose intolerance, Prader-Willi syndrome, HIV, cancer, renal failure, or cerebral palsy.
* They have tattoos, permanent makeup, dental ware, pacemakers, or metal implants that would preclude safe completion of the MRI.
* They have received an X-ray in the previous month.
* Their BMI-for-age percentile is between 85-95th

Parents :

* The biological mother has a body mass index < 18.5 kg/m2 or between 25-29.9 kg/m2.
* The primary parent in charge of making feeding decisions is unable to attend the study visits.
* The family reports plans to move away from the area in the next year.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
fMRI Neural Response to Food Portion Size Images | Baseline
  Functional magnetic resonance imaging (fMRI) will be used to measure brain activation in response to images of palatable, energy-dense food portions of varying sizes. Activation will be assessed in brain regions involved in visceral interoception (e.g., insula, cerebellum) and self-regulation (e.g., dorsolateral prefrontal cortex). These neural responses will be correlated with children's PACE phenotype scores to explore neurobiological underpinnings of eating behaviors.
PACE (Portion Size Susceptibility, Appetite Awareness, Loss of Control Eating, and Eating Speed) Phenotype Score | Baseline and 12-month follow-up
  The PACE score will be calculated as a composite measure including: 1) children's food intake during two laboratory meals with varying portion sizes, 2) parent-reported appetite traits via the Children's Eating Behavior Questionnaire, 3) loss of control eating measured with the Pediatric Eating Disorder Screener, and 4) eating rate quantified through video-recorded meals and behavioral coding of bite rate and eating speed. This score reflects obesogenic eating phenotypes.
Child Adiposity | Baseline and 12-month follow-up
  Child body fat percentage and adiposity will be measured using DXA scans, a validated imaging technique providing precise assessment of body composition. This measure will serve as the primary dependent variable to evaluate associations with PACE phenotype and changes over time.
Family Socioeconomic Status (SES) | Baseline
  Family SES will be assessed via parent self-report questionnaires, including family income levels and parental educational attainment. SES will be analyzed as a moderator of the relationship between PACE scores and child adiposity to explore social determinants of obesity risk.
PACE Phenotype Score Consistency Over Time | Baseline and 12-month follow-up
  PACE scores obtained at baseline and 12-month follow-up will be compared to evaluate the stability and trajectory of obesogenic eating behaviors in children over one year.

SECONDARY OUTCOMES:
Parent-reported race and ethnicity | Baseline
  Parent-reported information on the child's race and ethnicity collected via standardized questionnaire to capture demographic diversity and potential confounding factors.
Parent-reported socioeconomic status | Baseline
  Highest level of education completed by parents, self-reported, to help understand socioeconomic context and potential impact on child health and behavior.
Parent-reported educational attainment | Baseline
  Highest level of education completed by parents, self-reported, to help understand socioeconomic context and potential impact on child health and behavior.
Food security status | Baseline
  Parent-reported assessment of food security in the household using a validated food security questionnaire, to examine potential impact on child eating behaviors and adiposity.
Rurality of family home | Baseline
  Determined by family home zip code to classify rural versus urban residency, assessing environmental influences on child health and behavior.
Parent-reported feeding practices | Baseline
  Parent questionnaires assessing feeding styles, strategies, and control over child's food intake, providing insight into family eating environment.
Parent-reported appetitive traits | Baseline
  Parent assessment of child's appetite-related behaviors using standardized questionnaires to capture tendencies influencing eating patterns.
Child temperament | Baseline
  Parent-reported measures of child temperament characteristics to explore behavioral factors that might influence eating and activity.
Parent rating of child Tanner stage | Baseline
  Pubertal development stage assessed by parent report using Tanner scale, to account for physiological maturation impacting metabolism and behavior.
Child sleep patterns (parent-reported) | Baseline
  Parent-reported child sleep duration and quality via standardized sleep questionnaires to evaluate potential effects on weight and behavior.
Executive functioning | Baseline
  Direct child assessment of executive functions such as working memory, attention, and cognitive flexibility using the NIH Toolbox standardized tests.
Child IQ | Baseline
  Standardized assessment of child intelligence quotient using WASI-II.
Food liking and wanting during laboratory meals | Through study completion, an average of 1 year
  Child's hedonic ratings of food items consumed during laboratory meals to assess preferences influencing intake.
Food liking and wanting during fMRI scanning | Through study completion, an average of 1 year
  Child's ratings of liking and wanting for foods presented during fMRI scans to correlate brain activation with subjective food reward.
Pre-meal hunger and fullness ratings | Through study completion, an average of 1 year
  Child self-reported hunger and fullness before meals using visual analog scales to control for appetite state during intake measures.
Child visceral interoceptive awareness | Baseline
  Assessment of child's awareness of internal bodily signals via heartbeat perception task, indicating sensitivity to visceral cues potentially linked to eating behavior.
Child interoceptive awareness questionnaire | Baseline
  Child self-reported questionnaire measuring awareness of internal bodily sensations relevant to appetite and satiety.
Physical activity by accelerometry and questionnaire | Baseline
  Objective measurement of physical activity through accelerometer devices combined with parent and child questionnaires to quantify movement levels.
Sleep duration assessed by accelerometry | Baseline
  Sleep duration in hours per night
Intake at a standard baseline meal | Baseline
  Amount of food consumed by the child during a standardized meal in the laboratory setting to assess baseline intake independent of portion manipulation.
Intake of snacks and treats in the absence of hunger | Baseline
  Measurement of child's consumption of palatable snacks offered after a meal when not hungry, assessing loss of control or hedonic eating.
Relative reinforcing value of food assessed on computer task | Baseline
  Behavioral task evaluating the motivational value of food compared to alternative rewards, indicating reward sensitivity.
Sleep fragmentation index | Baseline
  Sleep fragmentation index is the number of 1 minute bouts of sleep divided by the total sleep time. Higher scores equal worse quality sleep.
Sleep Efficiency Percentage | Baseline
  Percent of time in bed that is spent asleep, with higher scores equal to better quality sleep.
Wake after sleep onset (WASO) | Baseline
  Minutes awake after onset of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Keller, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Metabolic Kitchen and Children's Eating Behavior Lab, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to PACE publication — https://pubmed.ncbi.nlm.nih.gov/38795747/